CLINICAL TRIAL: NCT06904547
Title: Resistance Mechanisms and Sequential Treatment Strategies Following First-Line Lorlatinib in ALK-Positive NSCLC: A Multi-center, Observational, Prospective Real-world Cohort Study (LORES)
Brief Title: Resistance Mechanisms and Sequential Treatment Strategies Following First-Line Lorlatinib in ALK-Positive NSCLC
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Ziming Li, Chief Physician, Shanghai Chest Hospital
Other Study IDs: IS25052
Record Dates: First submitted 2025-03-21; First posted 2025-04-01 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: ALK-Positive NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention administered — No intervention administered
Other: Non Interventional Study — Non Interventional Study

SUMMARY:
This is a prospective, multicenter, non-interventional, single-arm, real-world study planned to be conducted in China, aimed at exploring the resistance mechanisms of first-line lorlatinib treatment in patients with ALK-positive locally advanced or metastatic NSCLC, as well as the efficacy and safety of sequential treatments following lorlatinib resistance in the real-world setting.

ELIGIBILITY:
Inclusion Criteria

1. Age: Patients aged 18 years or older;
2. Histologically or cytologically confirmed locally advanced or metastatic NSCLC
3. Documened ALK resrrangemen by approved test (eg.. FisH,IHC. .r NGS).
4. first-line loelaninab treatment fom Apr2023-Apr-2027.
5. Evidenoe of popression to first-line lorlztinib within 2 weekes.

Exclusion Criteria

1. Previous treatment with other ALK-TKIs: Patients who have previously received any ALK TKI other than lorlatinib;
2. Concomitant medications: Patients who have received any systemic anti-tumor treatment other than lorlatinib before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with ALK-positive locally advanced or metastatic NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
mechanisms of resistance to first-line lorlatinib | 24 months
  Reslstance Assessment
  1. Liquld Blops-Blood eIDNA NGS
  2. Tissue Biopsy (If applicablo)-NGS
  mechanisms of resistance to first-line lorlatinib
  1. Propression pattern
     * Priary ressstance
     * Acquined resistance
  2. Moleculsr mechanisms of progression via ctDNA/organize NGS testing.
  3. Difference between the mnechsnisins of primary and acquired resistance

SECONDARY OUTCOMES:
Exploring the sequential treatment strategies and their efficacy and safety after first-line progression with lorlatinib | 24 months
  1. rwTTD1： discontinuation of lorlatinib for any reason (including disease progression, death, severe adverse events, or patient choice)
  2. rwTTD2： progression on first-line lorlatinib to discontinuation of the first sequential anti-tumor treatment for any reason (including disease progression, death, severe adverse events, or patient withdrawal from the study)
  3. rwORR2: the overall proportion of patients who achieve complete response (CR) and partial response (PR)
  4. rwDCR2: the overall proportion of patients who achieve complete response (CR), partial response (PR), and stable disease (SD)
  5. rwPFS2: progression on first-line lorlatinib to disease progression or death from any cause or last confirmed survival 6、1-year/2-year-rwPFS2 rate: he proportion of patients who remain progression-free within 1 year/2 years
  7、the overall proportion of patients who survive within 1 year/2 years 8、Exploration of the proportion and related reasons for dose adjustment

OTHER OUTCOMES:
To determine the optimal sequential treatment strategies for different resistance mechanisms and the impact of these resistance mechanisms on patient outcomes in sequential treatment | 24 months
  1. Explore the impact of different resistance mechanisms on patient prognosis, and investigate the sequential treatment strategies (including treatment efficacy and safety, if data are available in clinical practice) for ALK-positive locally advanced or metastatic NSCLC patients after resistance to first-line lorlatinib.
  2. Through comprehensive genomic analysis, explore which molecular pathological changes can provide guiding information for treatment after lorlatinib resistance, and identify which biomarkers can predict which patients are likely to benefit from specific treatments, thereby formulating individualized treatment plans to improve overall patient efficacy.